CLINICAL TRIAL: NCT02051595
Title: The Effects of Modified Ultrafiltration on Vancomycin Levels During Cardiopulmonary Bypass in Cardiac Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201300857
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Results first posted 2015-07-21 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Infection
Keywords: heart lung machine; blood pump; cardiac surgery; cardiopulmonary bypass; circulation
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vancomycin concentrations (Other): Up to ten blood samples testing for vancomycin concentrations will be collected in subjects administered vancomycin as prophylaxis before cardiac surgery with cardiopulmonary bypass and modified ultrafiltration.
  Interventions: Other: Vancomycin concentrations

INTERVENTIONS:
Other: Vancomycin concentrations — Up to ten blood samples testing for vancomycin concentrations will be collected in subjects administered vancomycin as prophylaxis before cardiac surgery with cardiopulmonary bypass and modified ultrafiltration.
  Other Names: pharmacodynamics; vancomycin monitoring; serum concentrations of vancomycin

SUMMARY:
Antibiotics are routinely used to prevent surgical wound infection. Vancomycin is a widely used antibiotic for surgery in patients with an allergy to penicillin. During cardiac surgery, cardiopulmonary bypass (CPB) and modified ultrafiltration (MUF) are routinely used and can lower the level of the antibiotic. The purpose of this study is to quantify the change in plasma vancomycin concentration associated with cardiopulmonary bypass and modified ultrafiltration.

DETAILED DESCRIPTION:
Subjects having cardiac surgery in which they will be on a heart-lung machine and will receive the antibiotic vancomycin, will be able to participate.

Up to ten blood samples testing for vancomycin concentrations will be collected in subjects administered vancomycin as prophylaxis before cardiac surgery with cardiopulmonary bypass and modified ultrafiltration. Participation will be complete once the cardiac surgery has been finished.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo cardiac surgery with cardiopulmonary bypass and modified ultrafiltration
* age greater than 18 years old
* penicillin allergy or in-hospital stay greater than 24 hours
* normal renal function
* normal liver function
* absence of clinical and laboratory signs of infection

Exclusion Criteria:

* vancomycin allergy
* pregnancy
* impaired renal function
* impaired liver function
* morbid obesity
* active infections
* Jehovah's Witness

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ettore Crimi, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vancomycin Concentrations: Vancomycin concentrations will be collected in subjects who are to undergo cardiac surgery with cardiopulmonary bypass and modified ultrafiltration.
  Vancomycin concentrations: Vancomycin concentrations will be collected in subjects who are to undergo cardiac surgery with cardiopulmonary bypass and modified ultrafiltration.
Period: Overall Study
Arm/Group | Vancomycin Concentrations
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vancomycin Concentrations
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Circulating Vancomycin Concentration
Description: Blood samples to monitor the vancomycin concentration will be collected at several time points during surgery.
Time Frame: Time points: pre CPB (t=1), post CPB at 5 (t=2), 30 (t=3), 60 (t=4), 108 (t=5), 240 (t=6) minutes, prior to ultrafiltration (t=7), end of ultrafiltration (t=8), ultrafiltrate (t=9) ,effluent of cell saver (t=10)
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Vancomycin Concentrations
Number analyzed (Participants) | 25
µg/mL | 15.6 (4.4)
Statistical Analysis 1: Comparison: Vancomycin Concentrations; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — A priori threshold was set to p < 0.05; Analyses modeled change in vancomycin concentrations (independent variable defined by time). Analyses were adjusted for covariates; estimate (beta) from mixed model = -0.068, 95% CI 2-sided [-0.098 to -0.039], Standard Error of Mean 0.015 — Negative beta value indicates that vancomycin concentration decreased following cardiopulmonary bypass (CPB)

ADVERSE EVENTS:
Time Frame: 12 hours
Arm/Group | Vancomycin Concentrations
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes